CLINICAL TRIAL: NCT02929693
Title: Clinical Study of Yiqi-yangyin-jiedu Decoction Combined With Gefitinib in Advanced Pulmonary Adenocarcinoma Patients With Activating EGFR Mutation
Brief Title: Clinical Study of YYJD Decoction Combined With Gefitinib in Advanced Pulmonary Adenocarcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Shanghai Chest Hospital (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Ling Xu, Principal Investigator, Shanghai University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHUTCM
Record Dates: First submitted 2016-10-08; First posted 2016-10-11 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- combination (Experimental): YYJD plus gefitinib
  Interventions: Drug: gefitinib; Drug: Yiqi-yangyin-jiedu decoction
- controll (Placebo Comparator): placebo plus gefitinib
  Interventions: Drug: gefitinib; Drug: placebo

INTERVENTIONS:
Drug: gefitinib — 250 mg oral once a day until progression or unacceptable toxicity develops
  Other Names: Iressa
Drug: Yiqi-yangyin-jiedu decoction — Yiqi-yangyin-jiedu decoction is a traditional chinese herbal medicine formula,and should be taken one package, twice a day, until progression or unacceptable toxicity develops.
  Other Names: YYJD
  Arms: combination
Drug: placebo — Oral granules, which the taste and smell are similar to YYJD, has no therapeutic effect, Oral granules, which the taste and smell are similar to experimental TCM granules, has no therapeutic effect, one package, twice a day, until progression or unacceptable toxicity develops.
  Other Names: control
  Arms: controll

SUMMARY:
The investigators performed a multi-centered, randomized, double blinded, placebo-controlled, prospective clinical trial on the effect of Yiqi-yangyin-jiedu decoction (YYJD), a chinese herbal medicine (CHM) formula combined with gefitinib to prolong the progression free survival (PFS) of advanced pulmonary adenocarcinoma patients with activating EGFR mutation (exon19del or exon21L858R). The investigators plan to enroll 198 cases in 3 years (99 cases for gefitinib, 99 cases for gefitinib plus YYJD), expecting that combination therapy has a better efficacy on prolonging PFS, overall survival, improving quality of life(QOL).

DETAILED DESCRIPTION:
Non-Small-Cell Lung Cancer（NSCLC）is one of the malignancies with high incidence and mortality. Epidermal growth factor receptor (EGFR) is implicated in NSCLC pathogenesis. Certain patient subgroups with NSCLC (ie, women, never-smokers, East Asians,adenocarcinoma) have higher rates of EGFR mutations, rendering them more responsive to EGFR tyrosine kinase inhibitors (TKIs; eg, gefitinib, erlotinib, Icotinib). Among patients with advanced EGFR-mutated NSCLC, treatment with EGFR-TKIs is associated with response rates of 56 to 74% and a median progression-free survival(mPFS) of 10 to 14 months;both outcomes are superior to those with platinum-based chemotherapy. Despite initial responses to EGFR-TKIs, the majority of patients will have disease progression within 1 to 2 years after treatment initiation (acquired resistance). In approximately 60% of patients, the mechanism of acquired resistance is the development of an additional EGFR mutation, EGFR T790M. Although AZD9291 (AstraZeneca), a third-generation EGFR-TKI is reported with a response rate of 61% in NSCLC patients with EGFR T790M and a mPFS of 9.6 months, resistance to third-generation inhibitors mediated by EGFR C797S mutation is inevitable. Therefore, optimizing the effect of each generation of EGFR-TKI is essential for long-term survival of NSCLC.The investigators' preliminary studies have shown that combining Yiqi-yangyin-jiedu decoction (YYJD) with gefitinib can prolong PFS and improve QOL, but high-level evidences are needed.

The investigators performed a multi-centered, randomized, double blinded, placebo-controlled, prospective clinical trial on the effect of YYJD, a chinese herbal medicine (CHM) formula combined with gefitinib in advanced pulmonary adenocarcinoma patients with activating EGFR mutation (exon19del or exon21L858R) that choose gefitinib as first-line or second line therapy. Patients are randomized into observational group (YYJD plus gefitinib),and control group (placebo plus gefitinib). The treatment should be continued until evidence of disease progression or unacceptable toxicity, and after that regular follow-up will be arranged. The primary efficacy assessments are: PFS (progression-free survival); Secondary efficacy assessments are: (1) OS (overall survival); (2) Objective response rate; (3) QOL (Functional Assessment of Cancer therapy-lung, FACT-L4.0 scales; Lung Cancer Symptom Scale, LCSS); (4) other efficacy assessments are: 1) TCM symptoms changes; 2) Toxicity, side effects and security of the treatments will be assessed at the same time. The investigators plan to enroll 198 cases in 3 years (99 cases for gefitinib, 99 cases for gefitinib plus YYJD), expecting that combination therapy has a better efficacy on prolonging PFS, overall survival, improving quality of life(QOL). Therefore the study can provide evidences for optimizing and promoting the efficacy of gefitinib.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or cytologically confirmed stage IIIa-IV pulmonary adenocarcinoma;
* With activating EGFR mutation (either exon19del or exon21L858R) and one month of gefitinib as first-line or second-line therapy without disease progression (PD);
* With TCM diagnostic pattern Qin-and-yin dificiency;
* Age ≥18 years old;
* Estimated life expectancy of at least 12 weeks;
* Without major organ dysfunction: hemoglobin ≥9 g/dL, absolute neutrophil count (ANC) ≥1.5*109/L, platelets ≥100 *109/L,bilirubin ≤1.5ULN, alkaline phosphatase (AP), aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 upper limited number(ULN) (AP, AST, ALT ≤5ULN is acceptable with liver metastasis).INR≤1.5, APTT in the normal range( 1.2DLN-1.2ULN),creatinine ≤1.5ULN;

Exclusion Criteria:

* with other malignant tumor except NSCLC 5 years previous to study entry;
* PD after onee month of gefitinib treatment
* Estimated life expectancy less than 12 weeks;
* Brain metastasis with relevant symptoms
* History of cardiovascular disease: Congestive Heart Failure > grade II in NYHA.Unstable angina patients (have angina symptoms in rest) or a new occurrence of angina (began in the last 3 months) or myocardial infarction happens in the last 6 months;
* Pregnant or child breast feeding women;

  * Mental or cognitive disorders;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 2 months
  Time from start of the study treatment to date of objective tumour progression (excluding clinical deterioration without evidence of objective progression).

SECONDARY OUTCOMES:
Overall survival (OS) | 2 months
  interval time from the first date of randomization to that of death for any reason, the end of the study, or loss of follow-up
Objective response rate (ORR) | 2 months
  The ORR (complete response (CR) plus partial response (PR)) was determined by the Response Evaluation Criteria In Solid Tumors (RECIST) (Eisenhauer et al, 2009) version 1.1.in Solid Tumors (RECIST1.1).
Quality of life (QOL) | 2 months
  QOL is assessed using Functional Assessment of Cancer therapy-lung (FACT-L) questionnaire .
Safety assessment evaluated according to Common Toxicity Criteria | 2 months
  Safety assessment is evaluated according to Common Toxicity Criteria (CTC 3.0).

IPD SHARING:
Plan to Share IPD: No